CLINICAL TRIAL: NCT05079906
Title: Assessment of Superficial Femoral Artery Lesions With FFR From the ACIST Navvus® Catheter
Acronym: FLO THRU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to timing
Sponsor: Acist Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US102
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Arterial Disease; Superficial Femoral Artery Stenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Main study arm (Other): All subjects will have their SFA lesion assessed with FFR measurement.
  Interventions: Device: Fractional Flow Reserve (FFR)
- Sub-study (Other): Last 50 enrolled subjects will have HD-IVUS in addition to FFR.
  Interventions: Device: Fractional Flow Reserve (FFR); Device: High Definition Intravascular Ultrasound (HD-IVUS)

INTERVENTIONS:
Device: Fractional Flow Reserve (FFR) — Fractional Flow Reserve (FFR) for all enrolled subjects. All interventional procedures, including FFR and HD IVUS, will be conducted in accordance with current approved User Guides and Instructions for Use.
Device: High Definition Intravascular Ultrasound (HD-IVUS) — High Definition Intravascular Ultrasound (HD-IVUS) in addition to FFR for last 50 enrolled subjects. All interventional procedures, including FFR and HD IVUS, will be conducted in accordance with current approved User Guides and Instructions for Use.
  Arms: Sub-study

SUMMARY:
This study is intended to help establish standard procedures for use of FFR in the peripheral arterial system and to evaluate the correlation of post-procedural FFR values and clinical outcomes in Superficial Femoral artery (SFA) interventions in subjects ages 18 to 79 with PAD.

DETAILED DESCRIPTION:
The ACIST Navvus Rapid Exchange FFR MicroCatheter is a rapid exchange catheter with a pressure sensor located at the distal tip that allows the operator to use their preferred standard 0.014-inch coronary guidewire for peripheral vascular intervention (PVI), eliminating the need for a wire exchange. The fractional flow reserve (FFR) measurements obtained with Navvus represent the degree of stenosis in an artery via comparison of the distal lesion value to the proximal lesion value.

While FFR has evolved as the gold standard for identifying coronary stenoses that may cause myocardial ischemia, it remains underutilized in the diagnosis and treatment of peripheral lesions. FFR cutoff values which could guide PVI decisions are yet to be defined and accepted. Routine use of FFR in patients with peripheral artery disease (PAD) may play an important role in determining the appropriateness of interventions in the peripheral vasculature by introducing a more objective assessment. Shishehbor and Agarwal further highlighted the potential economic benefit of FFR use in peripheral vessels by stating "The Affordable Care Act and higher emphasis on quality rather than quantity should support the use of [IVUS or FFR] to make peripheral interventions more accurate, safer, and better".

This study is intended to help establish standard procedures for use of FFR in the peripheral arterial system and to evaluate the correlation of post-procedural FFR values and clinical outcomes in Superficial Femoral artery (SFA) interventions in subjects ages 18 to 79 with PAD (Rutherford Classification 2, 3, 4, or 5). FFR measurements will be collected using the Navvus catheter pre- and post-PVI. A subset of study subjects will also have post-intervention IVUS imaging performed with the Kodama catheter.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79 at the time of planned SFA intervention
* SFA lesion requires intervention (according to ACC/AHA/SCAI/SIR/SVM 2018 Appropriate Use Criteria for Peripheral Artery Intervention, ABI, imaging, and/or clinical symptoms)
* Index SFA lesion is ≤150 mm
* Rutherford Classification of Peripheral Artery Disease (PAD) is Class 2, 3, 4, or 5
* Minimum two vessel run-off without a hemodynamically significant lesion below the treatment lesion (in at least one vessel to the foot) in the opinion of the treating physician

Exclusion Criteria:

* Study lesion is a Chronic Total Occlusion (CTO)
* Clinically significant (in the opinion of the treating physician) inflow disease of the aorta, common iliac, external iliac, or common femoral artery
* Presence of an additional hemodynamically significant stenosis within the SFA in the opinion of the treating physician
* Active cancer (any type)
* Life expectancy less than 1 year
* Pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Post-PVI FFR | 6 months
  Explore the correlation of post-PVI FFR values with other established clinical measures (i.e. 6MWT, ABI, VQ-6, WIQ, and arterial duplex US)

IPD SHARING:
Plan to Share IPD: No